CLINICAL TRIAL: NCT00916292
Title: A Phase 1a, Open Label, Single Dose, Dose Response, Pilot Study to Evaluate the Safety and Tolerability of Human Fibroblast Growth Factor-1 (FGF-1) in Normal Volunteers Given Punch Skin Biopsies
Brief Title: Safety Study of Topical Human FGF-1 for Wound Healing
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phage Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phage-W2009-01-1a
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes; dermal ulcers
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental): Four subjects will receive low dose FGF-1
  Interventions: Drug: FGF-1 141
- High Dose (Experimental): Four subjects will receive high dose FGF-1
  Interventions: Drug: FGF-1 141

INTERVENTIONS:
Drug: FGF-1 141 — Each subject will receive two, 3 mm squared punch skin biopsies, one biopsy will receive the study drug, and the second biopsy will remain untreated as a control. Low dose: FGF-1, 0.3 mg per square centimeter.
  Arms: Low dose
Drug: FGF-1 141 — Each subject will receive two, 3 mm squared punch skin biopsies, one biopsy will receive the study drug, and the second biopsy will remain untreated as a control. High dose: FGF-1, 3.0 mg per square centimeter.
  Arms: High Dose

SUMMARY:
The purpose of the study is to see if FGF-1 is safe when applied topically to the surface of a wound.

DETAILED DESCRIPTION:
Dermal ulcers pose a significant healthcare problem in the United States, ultimately affecting 10-15% of the approximately 20 million patients with diabetes and a similar number of patients with chronic venous insufficiency. Dermal leg and foot ulcers can result from compromised arterial inflow, microvascular perfusion or venous outflow which can lead to amputation unless vascular perfusion is improved. FGF-1 for topical administration offers the possibility of improved microvascular perfusion by promoting the formation of new blood vessels in the wound bed resulting in enhanced development of granulation tissue and accelerated healing.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form prior to the initiation of any study procedures. Subjects must be competent to give written informed consent.
2. Age must be between 18 to 75 years of age.
3. Female subject must be post-menopausal or sterilized, or if she is of childbearing potential, she is not breast feeding, and her serum pregnancy test is negative.
4. Subjects must be willing to change their wound dressings daily and demonstrate to study personnel the ability to follow the dressing care instructions indicated in the Appendix. Subjects considered eligible to enter the study must sign an informed consent form prior to the initiation of any study procedures. In the event that the subject must be withdrawn and is re-screened for study participation at a later date, a new informed consent form must be signed. Subjects must be competent to give written informed consent.

Exclusion Criteria:

1. Subjects receiving radiation therapy, corticosteroids, immunosuppressive agents or chemotherapy.
2. Subjects who, at study entry, are taking systemic antibiotics.
3. Subjects who are immunosuppressed.
4. Subjects experiencing bacterial or viral infection or who may otherwise be febrile.
5. Past history or current presence of any type of cancer (except past history of basal cell carcinoma that is not on the limb being treated). Subjects with existing BCC will be excluded from the study.
6. Life expectancy of less than 1 year.
7. Active alcohol or drug abuse within 6 months prior to study entry.
8. Screening liver function tests of more than 2.0 times the upper limit of normal.
9. Serum creatinine of ≥ 2.5 mg/dl.
10. Hemoglobin A1c (HgbA1c) of >10%.
11. Exposure to any other investigational drugs or devices or participation in any other investigational studies within 30 days prior to study entry.
12. Any other medical, social, or geographical factor that would make it unlikely that the subject will comply with study procedures (e.g., alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or a history of non-compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a single dose of FGF-1 topically administered in normal volunteers given an artificial dermal wound | 1 week

SECONDARY OUTCOMES:
Serum levels of FGF-1 after topical administration | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searle, MD, Principal Investigator — Dedicated Phase I
Locations (1):
- Dedicated Phase I, Phoenix, Arizona, United States